CLINICAL TRIAL: NCT01517399
Title: A Phase 1, Open-Label, Single-Sequence Crossover Study Assessing the Effect of Tivantinib (ARQ 197) on the Pharmacokinetics of Omeprazole/S-Warfarin/Caffeine/Midazolam and Digoxin in Cancer Subjects
Brief Title: Drug-drug Interaction Study of Tivantinib (ARQ 197) With Omeprazole, S-warfarin, Caffeine, Midazolam, and Digoxin in Cancer Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ARQ197-A-U158
Record Dates: First submitted 2012-01-04; First posted 2012-01-25 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2018-02

CONDITIONS: Solid Tumors
Keywords: Oncology; pharmacokinetics; PK interaction in advanced solid tumors with our drug and other drugs
MeSH Terms: conditions — Neoplasms | interventions — ARQ 197; Omeprazole; Warfarin; Caffeine; Vitamin K; Digoxin; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Test drug administration (Other): All drugs except vitamin K will be administered as a single dose once by itself as a reference treatment and once with tivantinib
  Interventions: Drug: tivantinib; Drug: omeprazole; Drug: s-warfarin; Drug: caffeine; Dietary Supplement: vitamin K; Drug: digoxin; Drug: midazolam

INTERVENTIONS:
Drug: tivantinib — three oral 120 mg tablets administered twice a day
  Other Names: ARQ 197
Drug: omeprazole — One 40 mg oral capsule once alone and once again with tivantinib
Drug: s-warfarin — One 10 mg oral tablet once alone and once again with tivantinib
Drug: caffeine — One 200 mg oral tablet once alone and once again with tivantinib
Dietary Supplement: vitamin K — One oral 5 mg tablet on multiple days when and around warfarin administration
Drug: digoxin — One oral 0.25 mg tablet once alone and once again with tivantinib
Drug: midazolam — Intravenous 1.5 mg dose once alone and once again with tivantinib

SUMMARY:
The purpose of this study is to determine the effects of tivantinib on the pharmacokinetics of omeprazole, s-warfarin, caffein, midazolam, or digoxin in patients with cancer.

DETAILED DESCRIPTION:
Nonclinical studies have indicated that tivantinib (parent molecule) has the potential to inhibit CYP3A4 ([I]/Ki=0.15, midazolam as substrate), CYP2C19 ([I]/Ki=0.98), CYP2C9 ([I]/Ki=0.44), and CYP1A ([I]/Ki=0.37), and the efflux transporter P glycoprotein (P-gp) (I2/IC50=82) at the clinical concentrations being studied in the Phase 3 development program. In addition, tivantinib has major circulating plasma metabolite(s) which also have been shown in nonclinical studies to exhibit similar CYP inhibition potential. The results of this study will evaluate the potential of tivantinib to influence the pharmacokinetics of CYP3A4/CYP2C19/CYP2C9/CYP1A and/or P-gp substrates, and help to provide the guidance to clinicians on co-administration of tivantinib with drugs metabolized by CYP3A4/CYP2C19/CYP2C9/ CYP1A and/or transported by P-gp.

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically or cytologically confirmed advanced solid tumor at screening;
2. Male or female ≥ 18 years of age;
3. Subjects (male and female) of childbearing potential must agree to use double barrier contraceptive measures or avoid intercourse during the study and for 90 days after the last dose of study drug. In addition, all female subjects of childbearing potential must have a negative pregnancy test result before initiating study treatment;
4. An Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
5. Adequate bone marrow, liver, clotting, and renal function, defined as:

   Platelet count ≥ 100 x 10^9/L, Hemoglobin (Hb) ≥ 9.0 g/dL, ANC ≥ 1.5 × 109/L, Total bilirubin ≤ 1.5 x the upper limit of normal (ULN), Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN (≤ 5 x ULN for subjects with liver metastases), International normalized ratio ≤ 1.5, Serum creatinine ≤ 1.5 x ULN;
6. Able to provide written informed consent, comply with protocol visits and procedures, be able to take oral medication, and not have any active infection or chronic co-morbidity that would interfere with therapy; and
7. Subjects must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects) and must sign and date an IRB approved ICF (including HIPAA authorization, if applicable) before performance of any study specific procedures or tests.

Exclusion Criteria:

1. History of cardiac disease:

   * Active coronary artery disease, defined as myocardial infarction (MI), unstable angina, coronary artery bypass graft, or stenting within 6 months prior to study entry (an MI that occurred > 6 months prior to study entry is permitted);
   * Evidence of uncontrolled symptomatic bradycardia or other cardiac arrhythmia defined as ≥ Grade 2 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4, or uncontrolled hypertension;
2. Active, clinically serious infection(s) defined as ≥ Grade 2 according to NCI CTCAE, version 4;
3. Family or personal history of coagulopathy;
4. History of hypersensitivity or adverse reactions to omeprazole, digoxin, warfarin, caffeine, midazolam, or vitamin K;
5. Known metastatic brain or meningeal tumors, unless the subject is > 3 months from definitive therapy and clinically stable (supportive therapy with steroids or anticonvulsant medications is allowed) with respect to the tumor at the time of first dose of study drug;
6. Pregnant or breastfeeding;
7. Any major surgical procedure within 3 weeks prior to first dose of study drug;
8. Significant gastrointestinal disorder(s), in the opinion of the Investigator (eg, Crohn's disease, ulcerative colitis, extensive gastric resection);
9. Received anti-cancer therapy, including antibody, retinoid, or hormonal treatment (except megestrol acetate as supportive care), and radiation, within 3 weeks before dosing. Prior and concurrent use of hormone replacement therapy, the use of gonadotropin-releasing hormone modulators for prostate cancer, and the use of somatostatin analogs for neuroendocrine tumors are permitted;
10. Received any other investigational drug within 3 weeks prior to dosing;
11. Received tivantinib as prior therapy;
12. Substance abuse or medical, psychological, or social conditions that may, in the opinion of the Investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results;
13. Any condition that is unstable or that could jeopardize the safety of the subject and the subject's protocol compliance, including known human immunodeficiency virus, hepatitis B virus, or hepatitis C virus infection;
14. Inability to swallow oral medications that could interfere with the absorption of tivantinib;
15. Administration or possibility of initiating or continuing any treatment with any known Cytochrome P450 (CYP)3A4, CYP2C19, CYP1A2, CYP2C9, and P-glycoprotein enzyme-altering drugs (inducer or inhibitor) or non-drug agents or systemic gastric pH modifiers (ie, ranitidine, proton pump inhibitors etc) within the 14 days prior to dosing and/or during the primary objective phase after initiation of the study treatment; or
16. Clinical diagnosis of hepatic impairment from chronic liver cirrhosis with confirmation by either previous liver biopsy or imaging, regardless of liver function test results at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-12; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) for S-Warfarin, Caffeine, Midazolam and Digoxin | Pharmacokinetic sampling will be done on days 1, 4, 6, 10, 11, 14, 16 (designated as days -5, -2, 1, 5, 6, 9, 11 in the study protocol)
  Parameters of S-warfarin/caffeine/midazolam and digoxin (area under the concentration-time curve from time 0 to the last quantifiable concentration [AUC last] and area under the curve from time of dosing extrapolated to infinity [AUC 0-inf]) when warfarin/caffeine/midazolam and digoxin are administered alone or in combination with tivantinib
Area under the plasma concentration versus time curve (AUC) for Omeprazole | Pharmacokinetic sampling will be done on days 1, 4, 6, 10, 11, 14, 16 (designated as days -5, -2, 1, 5, 6, 9, 11 in the study protocol)
  The ratios of omeprazole exposures vs. 5-hydroxyomeprazole exposures in terms of AUC last and AUC 0-inf when omeprazole is administered alone or in combination with tivantinib.

SECONDARY OUTCOMES:
Maximum observed concentration in plasma [Cmax] - Omeprazole, S-warfarin, Caffeine, Midazolam, Digoxin and the metabolite 5-hydroxyomeprazole | Pharmacokinetic sampling will be done on days 1, 4, 6, 10, 11, 14, 16 (designated as days -5, -2, 1, 5, 6, 9, 11 in the study protocol)
  Maximum observed concentration in plasma [Cmax] when omeprazole, warfarin, caffeine, midazolam and digoxin are administered alone or in combination with tivantinib.
Time to Maximum Plasma Concentration (Tmax) - Omeprazole, S-warfarin, Caffeine, Midazolam, Digoxin and the metabolite 5-hydroxyomeprazole | Pharmacokinetic sampling will be done on days 1, 4, 6, 10, 11, 14, 16 (designated as days -5, -2, 1, 5, 6, 9, 11 in the study protocol)
  Maximum observed concentration in plasma [Tmax] when omeprazole, warfarin, caffeine, midazolam and digoxin are administered alone or in combination with tivantinib.
Apparent oral clearance [CL/F] - Omeprazole, S-warfarin, Caffeine, Midazolam, Digoxin and the metabolite 5-hydroxyomeprazole | Pharmacokinetic sampling will be done on days 1, 4, 6, 10, 11, 14, 16 (designated as days -5, -2, 1, 5, 6, 9, 11 in the study protocol)
  Apparent oral clearance [CL/F] when omeprazole, warfarin, caffeine, midazolam and digoxin are administered alone or in combination with tivantinib.
Apparent volume of distribution [V/F] - Omeprazole, S-warfarin, Caffeine, Midazolam, Digoxin and the metabolite 5-hydroxyomeprazole | Pharmacokinetic sampling will be done on days 1, 4, 6, 10, 11, 14, 16 (designated as days -5, -2, 1, 5, 6, 9, 11 in the study protocol)
  Apparent volume of distribution [V/F] when omeprazole, warfarin, caffeine, midazolam and digoxin are administered alone or in combination with tivantinib.
Maximum observed concentration in plasma [Cmax] for Tivantinib and its major metabolites, HPM4, HPM5, HPM6, and HPM8 | Pharmacokinetic sampling will be done on Days 6, 10, and 16 (designated as days 1, 5, and 11 in the study protocol)
Time to Maximum Plasma Concentration (Tmax) for Tivantinib and its major metabolites, HPM4, HPM5, HPM6, and HPM8 | Pharmacokinetic sampling will be done on Days 6, 10, and 16 (designated as days 1, 5, and 11 in the study protocol)
Apparent oral clearance [CL/F] for Tivantinib and its major metabolites, HPM4, HPM5, HPM6, and HPM8 | Pharmacokinetic sampling will be done on Days 6, 10, and 16 (designated as days 1, 5, and 11 in the study protocol)
Apparent volume of distribution [V/F] for Tivantinib and its major metabolites, HPM4, HPM5, HPM6, and HPM8 | Pharmacokinetic sampling will be done on Days 6, 10, and 16 (designated as days 1, 5, and 11 in the study protocol)

CONTACTS AND LOCATIONS:
Overall Officials: Hamim Zahir, BPharm, PhD, Study Director — Daiichi Sankyo UK Ltd.
Locations (1):
- START - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/